CLINICAL TRIAL: NCT06429644
Title: Ong-term Oncologic Outcome of Breast-conserving Surgery in Breast Cancer Patients With BRCA1/2 Mutations
Brief Title: Long-term Oncologic Outcome of Breast-conserving Surgery in Breast Cancer Patients With BRCA1/2 Mutations
Status: Completed | Type: Observational
Sponsor: Hanyang University Seoul Hospital (Other)
Collaborators: Korean Surgical Society (Unknown); Korea Robot-Endoscopy Minimal Access Breast Surgery Study Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-04-039
Record Dates: First submitted 2024-04-30; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-04

CONDITIONS: BRCA1/2 Mutation; Breast-conserving Surgery
MeSH Terms: interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (13):
- Dongtan Sacred Heart Hospital: Department of Surgery, Dongtan Sacred Heart Hospital, Hallym University, Dongtan, Republic of Korea
  Interventions: Procedure: Breast-conserving surgery
- Samsung Medical Center: Division of Breast Surgery, Department of Surgery, Sungkyunkwan University School of Medicine, Samsung Medical Center, Seoul, Republic of Korea
  Interventions: Procedure: Breast-conserving surgery
- Seoul National University Hospital: Breast Care Center, Department of Surgery, Seoul National University Hospital, Seoul, Republic of Korea
  Interventions: Procedure: Breast-conserving surgery
- Severance hospital: Department of Surgery, Severance hospital, Yonsei University College of Medicine, Seoul, Republic of Korea
  Interventions: Procedure: Breast-conserving surgery
- Kyungpook National University Chilgok Hospital: Department of Surgery, School of Medicine, Kyungpook National University, Kyungpook National University Chilgok Hospital, Daegu, Republic of Korea
  Interventions: Procedure: Breast-conserving surgery
- Gangnam Severance Hospital: Department of Surgery, Gangnam Severance Hospital, Yonsei University College of Medicine, Seoul, Republic of Korea
  Interventions: Procedure: Breast-conserving surgery
- Hanyang University Medical Center: Department of Surgery, Hanyang University Medical Center, Hanyang University College of Medicine, Seoul, Republic of Korea
  Interventions: Procedure: Breast-conserving surgery
- Hallym University Sacred Heart Hospital: Department of Breast & Endocrine Surgery, Hallym University Sacred Heart Hospital, Hallym University, Anyang, Republic of Korea
  Interventions: Procedure: Breast-conserving surgery
- Kangbuk Samsung Hospital: Department of Surgery, Kangbuk Samsung Hospital, Sungkyunkwan University School of Medicine, Seoul, Republic of Korea
  Interventions: Procedure: Breast-conserving surgery
- Incheon St. Mary's Hospital: Department of Surgery, Incheon St. Mary's Hospital, College of Medicine, The Catholic University of Korea, Incheon, Republic of Korea
  Interventions: Procedure: Breast-conserving surgery
- Kyung Hee University Hospital: Department of Surgery, Kyung Hee University Hospital, Seoul, Republic of Korea
  Interventions: Procedure: Breast-conserving surgery
- Keimyung University School of Medicine: Department of Surgery, Keimyung University School of Medicine, Daegu, Republic of Korea
  Interventions: Procedure: Breast-conserving surgery
- Asan Medical Center: Division of Breast Surgery, Department of Surgery, University of Ulsan College of Medicine, Asan Medical Center, Seoul, Republic of Korea
  Interventions: Procedure: Breast-conserving surgery

INTERVENTIONS:
Procedure: Breast-conserving surgery — Breast-conserving surgery, also known as breast-conserving therapy or lumpectomy, is a surgical procedure used to treat breast cancer while preserving as much of the breast tissue as possible. During this procedure, the surgeon removes the cancerous tumor along with a surrounding margin of normal tissue. The goal is to remove the cancerous cells while maintaining the appearance and function of the breast as much as possible.

SUMMARY:
The investigators matched BCS and mastectomy group using propensity scores and analyzed the recurrence and survival among the evenly matched patients in breast cancer patients with BRCA 1/2 mutations.

DETAILED DESCRIPTION:
The purpose of study is to assess the oncologic safety of BCS in patients carrying BRCA1/2 mutations by comparing long-term outcomes with mastectomy. The investigators matched BCS and mastectomy group using propensity scores and analyzed the recurrence and survival among the evenly matched patients. By providing insights into the feasibility of BCS for patients with BRCA1/2 mutations, the investigators aim to present evidence to aid in surgical decision-making for the care of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary invasive breast cancer who underwent BCS or mastectomy
* Received a BRCA1/2 mutation test

Exclusion Criteria:

* Patients with de novo metastasis
* Pregnancy-associated breast cancer

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The ON-BRCAII is multi-institution cohort study being conducted by the Korea Robot-Endoscopy Minimal Access Breast Surgery Study Group (KoREa-BSG). Patients with primary breast cancer who underwent BCS or mastectomy and received a BRCA1/2 mutation test between January 2008 and December 2015 were retrospectively identified from 13 institutions in South Korea. The inclusion criteria comprised patients aged 20 to 80 years with invasive breast cancer (pT1-3, N0-3). The exclusion criteria consisted of patients with de novo metastasis and those with pregnancy-associated breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 4010 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Locoregional recurrence-free survival | Duration from diagnosis until the development of recurrence up to 10year
  Recurrence in breast or chest wall and/or regional lymph nodes
Distant recurrence-free survival | Duration from diagnosis until the development of recurrence up to 10year
  Recurrence in a distant organ
Recurrence-free survival | Duration from diagnosis until the development of recurrence up to 10year
  Any form of disease recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang university hospital, Seoul, South Korea